CLINICAL TRIAL: NCT06203587
Title: Clinical Study of GPA33-specific PET/CT for the Diagnosis of Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-1016
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Positron-Emission Tomography; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with colorectal cancer (Experimental): Subjects were recruited from the Department of Gastroenterology, Huashan Hospital, Fudan University, Shanghai, China.
  Interventions: Radiation: [68Ga]Ga-NOTA-WWH347 or [18F]F-H3RESCA-WWH347

INTERVENTIONS:
Radiation: [68Ga]Ga-NOTA-WWH347 or [18F]F-H3RESCA-WWH347 — The dose of [68Ga]Ga-NOTA-WWH347 or [18F]F-H3RESCA-WWH347, calculated from the patient's body weight, was 1.8-3.7 MBq [0.05-0.1 mCi]/kg, and was administered as an intravenous push, with a single dose given once.

SUMMARY:
In this study, we will first investigate the imaging safety and feasibility of [68Ga]Ga-NOTA-WWH347 and [18F]F-H3RESCA-WWH347 PET/CT in patients with primary and/or metastatic colorectal cancers. The second goal of the study is to preliminarily investigate the diagnostic efficacy (e.g., sensitivity and specificity) of [68Ga]Ga-NOTA-WWH347 and [18F]F-H3RESCA-WWH347 PET/CT in patients with primary and/or metastatic colorectal cancers. This study will provide a new method for the noninvasive target-specific diagnosis of colorectal cancer, and provide an intuitive and clear imaging basis for clinical diagnosis, differential diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 65 years of age and of either sex.
2. Patients with colorectal cancer confirmed by puncture or surgical pathology.
3. Written informed consent signed by the subject or legal guardian or caregiver.
4. Willingness and ability to cooperate with all programs of this study.

Exclusion Criteria:

1. Severe hepatic or renal insufficiency;
2. Targeted therapy before radiotherapy or PET/CT scan. Renal function: serum creatinine less than or equal to the upper limit of the normal range;
3. Liver function: bilirubin, AST(SGOT)/ALT(SGPT) less than or equal to the upper limit of the normal range.
4. History of serious surgery in the last month.
5. Those who have participated in other clinical trials during the same period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Establishment and optimization of imaging method for [68Ga]Ga-NOTA-WWH347 or [18F]F-H3RESCA-WWH347 PET/CT. | 90mins from time of injection
  To assess the safety, sensitivity and specificity of diagnosing colorectal cancer using [68Ga]Ga-NOTA-WWH347 or [18F]F-H3RESCA-WWH347 PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China